CLINICAL TRIAL: NCT00637546
Title: Efficacy of a Specific Physiotherapy Group Treatment on Gait and Balance in Patients With Diabetic Neuropathy
Brief Title: Gait and Balance of Diabetes Type 2 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Maastricht University Medical Center (Other); Swiss Federal Institute of Technology (Other); Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Lara Allet (Mrs), University Hopsital Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-305
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Type 2
Keywords: Treatment; Efficacy; Diabetes; Gait; Balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A,1 (Experimental): Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Gait and Balance training based on recommendations of Robertson et al. and Page et al. (different balance control exercises; progression in consecutive stages: Sensimotor training, a static phase, a dynamic phase combined with functional tasks. The treatment takes place twice a week over 12 weeks. Patients were encouraged to perform specific home exercises.
  Other Names: Physical Therapy

SUMMARY:
Type 2 diabetes is one of the fastest growing public health problems in both developed and developing countries. It is estimated that the number of people with diabetes in the world will double in coming years, from 171 million in 2000 to 366 million in 2030.The role of physiotherapy in diabetic care is to reduce immobilisation effects, to maintain functional capacity and to minimise diabetes-related complications. The physiotherapist also has a role in providing advice about exercise and daily living activities. The fundamental principle of rehabilitation is to improve quality of life while diminishing the health care burden. By reducing the heightened risk of falling, the fall related injuries and the fear of falling one could improve quality of life in diabetic patients and reduce health care costs.

The goal of this study is to investigate the effectiveness of gait and balance training in pre frail subgroup diabetes patients. Our program is based on recommendations of Robertson et al.(2002) and Page et al.(2002) The investigators randomly assign patients in a control group (no treatment) or in a treatment group. The treatment program consists of two group sessions per week over 12 weeks. Patients were encouraged to perform specific home exercises. After this 12-week program, patients were asked to continue their exercises. The effect of the treatment will be evaluated after the treatment program and after a 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Past or present patient from the University Hospital in Geneva
* Diagnosed with diabetes by the medical doctor (glycaemia > 7 mmol on two different tests on an empty stomach)
* Presence of a peripheral neuropathy (vibration perception ≤ 4)

Exclusion Criteria:

* Patients with a foot ulcer at the moment of intake
* Patients with orthopaedic or chirurgical problems influencing gait parameters
* Patients with a non diabetic neuropathy (Charcot, alcohol, Thyroid dysfunction)
* Patients with neurological problems influencing gait parameters
* Patients with incapacity to walk without a walking aid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Gait parameter: comfortable speed | Before treatment / After treatment / 6 month follow up

SECONDARY OUTCOMES:
Other spatio temporal gait parameters and sagittal movement of lower limb | Before Treatment/ After Treatment/ 6 month follow up
Balance measures (Tinetti and Biodex balance Index, acceleration on sacrum) | Before Treatment / After Treatment / 6 month follow up
Fear of falling (Falls efficacy scale) | Before Treatment / After Treatment / 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Lara E Allet, MPtSc, Principal Investigator — University Hospital and University Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Allet L, Armand S, Golay A, Monnin D, de Bie RA, de Bruin ED. Gait characteristics of diabetic patients: a systematic review. Diabetes Metab Res Rev. 2008 Mar-Apr;24(3):173-91. doi: 10.1002/dmrr.809. PMID 18232063
- [Background] Turcot K, Allet L, Golay A, Hoffmeyer P, Armand S. Investigation of standing balance in diabetic patients with and without peripheral neuropathy using accelerometers. Clin Biomech (Bristol). 2009 Nov;24(9):716-21. doi: 10.1016/j.clinbiomech.2009.07.003. Epub 2009 Aug 14. PMID 19683372
- [Result] Allet L, Armand S, de Bie RA, Golay A, Monnin D, Aminian K, Staal JB, de Bruin ED. The gait and balance of patients with diabetes can be improved: a randomised controlled trial. Diabetologia. 2010 Mar;53(3):458-66. doi: 10.1007/s00125-009-1592-4. Epub 2009 Nov 17. PMID 19921145
- [Result] Allet L, Armand S, de Bie RA, Golay A, Pataky Z, Aminian K, de Bruin ED. Clinical factors associated with gait alterations in diabetic patients. Diabet Med. 2009 Oct;26(10):1003-9. doi: 10.1111/j.1464-5491.2009.02811.x. PMID 19900232
- [Result] Allet L, Armand S, de Bie RA, Pataky Z, Aminian K, Herrmann FR, de Bruin ED. Gait alterations of diabetic patients while walking on different surfaces. Gait Posture. 2009 Apr;29(3):488-93. doi: 10.1016/j.gaitpost.2008.11.012. Epub 2009 Jan 9. PMID 19138520
- [Result] Allet L, Armand S, de Bie RA, Golay A, Monnin D, Aminian K, de Bruin ED. Reliability of diabetic patients' gait parameters in a challenging environment. Gait Posture. 2008 Nov;28(4):680-6. doi: 10.1016/j.gaitpost.2008.05.006. Epub 2008 Jun 25. PMID 18579384